CLINICAL TRIAL: NCT02407613
Title: Efficacy of Magnetic Resonance-guided High Intensity Focused Ultrasound for the Ablation of Breast Cancer
Brief Title: Efficacy of MR-HIFU Ablation of Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient recruitment was not feasible.
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Manon Braat, MD, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL46863.041.14
Record Dates: First submitted 2015-01-16; First posted 2015-04-03 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; MR-HIFU; ablation; non-invasive treatment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MR-HIFU ablation (Experimental): Ten patients undergo MR-HIFU ablation with the Sonalleve MR-HIFU Breast Tumor Therapy System (Profound Medical). According to a treat-and-resect protocol, these patients also undergo standard therapy consisting of breast cancer surgery 1 to 2 weeks after MR-HIFU treatment (+/- radiotherapy).
  Interventions: Device: Philips Sonalleve MR-HIFU Breast Tumor Therapy System

INTERVENTIONS:
Device: Philips Sonalleve MR-HIFU Breast Tumor Therapy System — Magnetic Resonance-guided High-Intensity Focused Ultrasound (MR-HIFU) is a completely non-invasive treatment technique. HIFU uses focused ultrasound to achieve temperature rise in the targeted tissue. Real time monitoring of the treatment with MR-thermometry is used to ensure optimal safety.

SUMMARY:
This study evaluates the efficacy of MR-HIFU ablation of breast cancer. Ten patients with early-stage breast cancer with a maximum diameter of 3 cm will undergo MR-HIFU ablation, followed by MRI and surgical resection to evaluate treatment effect. The main purpose of the study is to demonstrate the feasibility of total tumor ablation with MR-HIFU. The secondary objective is safety assessment.

ELIGIBILITY:
Inclusion Criteria:

* Women, aged 18 years and older.
* Able to give informed consent herself.
* World Health Organization (WHO) performance score ≤ 2.
* Biopsy proven cT1-2 N0-2 MX invasive breast cancer with a size of ≤ 3.0 cm.
* Histological type of tumor: invasive ductal carcinoma (IDC), not otherwise specified (NOS) or no special type (NST).
* The target breast fits in the cup of the dedicated MR-HIFU breast system.
* Patient weight is limited to ≤ 90 kg, because of restrictions to the HIFU table top.

Additional inclusion criteria based on DCE-MRI findings:

* The distance of the tumor, including a 5 mm margin around the tumor, from the skin, nipple and pectoral wall is at least 1.0 cm measured on MRI.
* The tumor is located within the reach of the HIFU beam produced by the transducers in the HIFU breast system.

Exclusion Criteria:

* Prior treatment with: neo-adjuvant systemic therapy in the past 3 months or radiotherapy or thermal therapy or surgery of any kind in the targeted breast.
* Contraindications to MR imaging according to the hospital guidelines (e.g. pacemaker in situ, severe claustrophobia, big metal implants, body size incompatible with MR bore).
* Contraindications to administration of gadolinium-based contrast agent, including: prior allergic reaction to a gadolinium-based contrast agent, kidney disease (e.g. nephrogenic systemic fibrosis, nephrogenic fibrosing dermopathy) and/or renal failure (GFR < 30 ml/min/1,73m2).
* Contra-indications for procedural sedation analgesia with Propofol and Esketamine or Propofol and Remifentanil.
* Extensive intraductal components in the lesion determined by biopsy.
* Scar tissue or surgical clips in the HIFU beam path.
* Inability to lie in prone position.
* Pregnancy or lactation.
* Communication barrier with patient.

The following groups of patients will be excluded because the risk of adjuvant over- or undertreatment due to performing the Bloom and Richardson (B&R) grading on the tumor biopsy is considered to high:

* N0, Her2neu negative, <35 years, ≤1cm (T1a/b) with B&R grade 1 or 2 on biopsy.
* N0 Her2neu negative, ER/PR negative (triple negative), 35-70yr, 1.1-2cm (T1c) with B&R grade 1 or 2 on biopsy.
* N0, Her2neu negative, ER/PR positive > 50%, ductal carcinoma, 60-70yr, 1.1-2cm (T1c), with B&R grade 3 on biopsy and if the MammaPrint is not reimbursed by health insurance also for grade 1 on biopsy.
* N0, Her2neu negative, ER/PR positive, ductal carcinoma, 35-60yr, 1.1-2cm (T1c) with B&R grade 1 on biopsy.
* N0, Her2neu negative, ER/PR positive, but ≤50%, ductal carcinoma, 60-70yr, 1.1-2cm (T1c) with B&R grade 1.

The following group of patients will be excluded based on the results of the MammaPrint:

• Only if the MammaPrint is reimbursed by health insurance: N0, Her2neu negative, ER/PR positive, > 50% ductal carcinoma, 60-70yr, 1.1-2cm (T1c), with B&R grade 1 and MammaPrint high risk.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Amount of ablated tissue at histopathological examination | 2-3 weeks (after surgery is performed)
  The amount of ablated tissue and residual viable tumor tissue will be assessed in all tumor slices.
Presence of non-perfused volumes on DCE-MRI | 1 week after MR-HIFU ablation
  Efficacy will be assessed by the presence of non-perfused volumes on DCE-MRI. A pre-treatment MRI is used as comparison.

SECONDARY OUTCOMES:
Number of patients with adverse events | Approximately 2 to 3 weeks
  Adverse events will be documented. The (possible) relationship with MR-HIFU ablation will be asessed in all cases.

CONTACTS AND LOCATIONS:
Overall Officials: Manon NG Braat, MD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands